CLINICAL TRIAL: NCT01863043
Title: Routine Aspiration of Residual Gastric Contents in Very Low Birth Weight Infants
Brief Title: Aspiration of Residual Gastric Contents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB201501174- N; 1R01NR014019-01A1 (NIH)
Record Dates: First submitted 2013-05-22; First posted 2013-05-27 (Estimated); Results first posted 2023-06-28 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Infant, Premature; Nutrition, Enteral
Keywords: Premature Infant; Nutrition; Enteral
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine aspiration of gastric contents (Active Comparator): Infants will have routine aspiration of gastric contents prior to each feeding to monitor the amount of residual gastric contents remaining in the stomach.
  Interventions: Procedure: Routine aspiration of gastric contents
- No aspiration of gastric contents (Experimental): Infants will not have routine aspiration of gastric contents prior to every feeding to assess residual gastric contents.
  Interventions: Procedure: No aspiration of gastric contents

INTERVENTIONS:
Procedure: No aspiration of gastric contents — Infants will not have routine aspiration of gastric contents prior to every feeding to assess residual gastric contents.
  Arms: No aspiration of gastric contents
Procedure: Routine aspiration of gastric contents — Infants will have routine aspiration of gastric contents prior to each feeding to monitor the amount of residual gastric contents remaining in the stomach.
  Arms: Routine aspiration of gastric contents

SUMMARY:
The primary purpose of this study is to determine nutrition outcomes and risks to gastrointestinal integrity and function of aspirating for routine gastric contents prior to each feeding in very low birth weight premature infants.

DETAILED DESCRIPTION:
The participants in the study will be randomly assigned (like the flip of a coin) to either have the leftover food in their stomach removed before each feeding, or not have the leftover food removed before each feeding. In addition, when a blood drawn is performed as regular care an extra amount with be taken. A test to determine how much of the hormones gastrin and motilin are contained in the blood will be performed. Stool samples will be collected. Participation could last up to approximately 6 to 8 weeks of age.

ELIGIBILITY:
Inclusion Criteria:

* born at 32 weeks of less of gestational age
* birth weight </= to 1250 grams
* receiving some enteral feedings by 72 hours of age
* receiving parenteral feedings by 24 hours of age

Exclusion Criteria:

* Congenital or chromosomal abnormalities
* complex congenital heart diseases and congenital anatomic gastrointestinal abnormalities

Max Age: 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 146 (Actual)
Dates: Start 2013-10-07 (Actual); Primary Completion 2016-10-08 (Actual); Study Completion 2019-01-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leslie A Parker, PhD, Principal Investigator — University of Florida
Locations (1):
- Neonatal intensive care unit at Shands children's hospital at the Univeristy of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Parker LA, Weaver M, Murgas Torrazza RJ, Shuster J, Li N, Krueger C, Neu J. Effect of Aspiration and Evaluation of Gastric Residuals on Intestinal Inflammation, Bleeding, and Gastrointestinal Peptide Level. J Pediatr. 2020 Feb;217:165-171.e2. doi: 10.1016/j.jpeds.2019.10.036. Epub 2019 Nov 19. PMID 31757473
- [Derived] Parker LA, Weaver M, Murgas Torrazza RJ, Shuster J, Li N, Krueger C, Neu J. Effect of Gastric Residual Evaluation on Enteral Intake in Extremely Preterm Infants: A Randomized Clinical Trial. JAMA Pediatr. 2019 Jun 1;173(6):534-543. doi: 10.1001/jamapediatrics.2019.0800. PMID 31034045

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred between 10/17/2013 and 10/8/2016 in a Level 4 neonatal intensive care unit
Pre-assignment Details: No participants were excluded before assignment to groups
Period: Overall Study
Arm/Group | Routine Aspiration of Gastric Contents | No Aspiration of Gastric Contents
Started | 74 | 72
Completed | 61 | 60
Not Completed | 13 | 12
Not completed — Death | 6 | 1
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Adverse Event | 7 | 8
Not completed — exclusion criteria found after enrollment | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Routine Aspiration of Gastric Contents | No Aspiration of Gastric Contents | Total
Number analyzed (Participants) | 74 | 72 | 146
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 74 | 72 | 146
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: weeks] — Gestational age at birth
  weeks | 27.1 (2.4) | 27 (1.2) | 27.03 (2.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 37 | 74
  Male | 37 | 35 | 72
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 22 | 42 | 64
  White | 49 | 28 | 77
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Enteral Intake on Day of Life 7
Description: The volume in mL/kg of feeds provided to infant on day of life 7
Time Frame: Day of life 7
Measure: Least Squares Mean (95% Confidence Interval); unit: mL/kg per day
Arm/Group | Routine Aspiration of Gastric Contents | No Aspiration of Gastric Contents
Number analyzed (Participants) | 74 | 69
mL/kg per day | 27.5 [21.8 to 29.5] | 22.6 [18.6 to 26.5]
Statistical Analysis 1: Comparison: Routine Aspiration of Gastric Contents vs No Aspiration of Gastric Contents; Test type: Superiority; p = 0.27, Mixed Models Analysis

2. Primary Outcome: Enteral Intake on Day of Life 14
Description: The volume in mL/kg of feeds provided to infant on day of life 7
Time Frame: Day of life 14
Measure: Least Squares Mean (95% Confidence Interval); unit: mL/kg per day
Arm/Group | Routine Aspiration of Gastric Contents | No Aspiration of Gastric Contents
Number analyzed (Participants) | 74 | 69
mL/kg per day | 83.2 [72.9 to 93.8] | 94.7 [84.3 to 105.2]
Statistical Analysis 1: Comparison: Routine Aspiration of Gastric Contents vs No Aspiration of Gastric Contents; Test type: Superiority; p = 0.12, Mixed Models Analysis

3. Primary Outcome: Enteral Intake on Day of Life 21
Description: The volume in mL/kg of feeds provided to infants on day of life 21
Time Frame: Day of life 21
Measure: Least Squares Mean (95% Confidence Interval); unit: mL/kg per day
Arm/Group | Routine Aspiration of Gastric Contents | No Aspiration of Gastric Contents
Number analyzed (Participants) | 74 | 69
mL/kg per day | 109.2 [98.5 to 120] | 117.7 [106.9 to 128.5]
Statistical Analysis 1: Comparison: Routine Aspiration of Gastric Contents vs No Aspiration of Gastric Contents; Test type: Superiority; p = 0.28, Mixed Models Analysis

4. Primary Outcome: Enteral Intake on Day of Life 28
Description: The volume in mL/kg of feeds provided to the infant on day of life 28
Time Frame: Day of life 28
Measure: Least Squares Mean (95% Confidence Interval); unit: mL/kg per day
Arm/Group | Routine Aspiration of Gastric Contents | No Aspiration of Gastric Contents
Number analyzed (Participants) | 74 | 69
mL/kg per day | 119.4 [109.5 to 129.6] | 129.6 [119.7 to 139.6]
Statistical Analysis 1: Comparison: Routine Aspiration of Gastric Contents vs No Aspiration of Gastric Contents; Test type: Superiority; p = 0.15, Mixed Models Analysis

5. Primary Outcome: Enteral Intake at Day of Life 35
Description: The volume in mL/kg of feeds provided to infants on day of life 35
Time Frame: Day of life 35
Measure: Least Squares Mean (95% Confidence Interval); unit: mL/kg per day
Arm/Group | Routine Aspiration of Gastric Contents | No Aspiration of Gastric Contents
Number analyzed (Participants) | 74 | 69
mL/kg per day | 123.9 [115.2 to 132.6] | 137.2 [128.6 to 145.8]
Statistical Analysis 1: Comparison: Routine Aspiration of Gastric Contents vs No Aspiration of Gastric Contents; Test type: Superiority; p = 0.03, Mixed Models Analysis

6. Primary Outcome: Enteral Intake on Day of Life 42
Description: The volume in mL/kg of feeds provided to infants on day of life 42
Time Frame: Day of life 42
Measure: Least Squares Mean (95% Confidence Interval); unit: mL/kg per day
Arm/Group | Routine Aspiration of Gastric Contents | No Aspiration of Gastric Contents
Number analyzed (Participants) | 74 | 69
mL/kg per day | 128.4 [119.9 to 136.9] | 141.6 [133.2 to 150]
Statistical Analysis 1: Comparison: Routine Aspiration of Gastric Contents vs No Aspiration of Gastric Contents; Test type: Superiority; p = 0.03, Mixed Models Analysis

7. Secondary Outcome: Days to Reach Full Feeds
Description: Full feeds is defined as 120 milliliters per kilogram per day
Time Frame: baseline to approximately 42 days
Measure: Least Squares Mean (95% Confidence Interval); unit: days
Arm/Group | Routine Aspiration of Gastric Contents | No Aspiration of Gastric Contents
Number analyzed (Participants) | 74 | 69
days | 18.1 [16.3 to 20] | 15.9 [14.1 to 17.8]
Statistical Analysis 1: Comparison: Routine Aspiration of Gastric Contents vs No Aspiration of Gastric Contents; Test type: Superiority; p = 0.59, Accelerated failure time regression mode

8. Secondary Outcome: Hours Receiving Parenteral Nutrition
Description: The number of hours participants required parenteral nutriton
Time Frame: Baseline to 42 days
Measure: Least Squares Mean (95% Confidence Interval); unit: hours
Arm/Group | Routine Aspiration of Gastric Contents | No Aspiration of Gastric Contents
Number analyzed (Participants) | 74 | 69
hours | 358.8 [312.2 to 405.4] | 356.8 [310.6 to 403.1]
Statistical Analysis 1: Comparison: Routine Aspiration of Gastric Contents vs No Aspiration of Gastric Contents; Test type: Superiority; p = 0.64, Accelerated failure time regression mode

9. Secondary Outcome: Hours of Central Line Access
Description: The number of hours participants required central line access
Time Frame: Baseline to 42 days
Measure: Least Squares Mean (95% Confidence Interval); unit: Hours
Arm/Group | Routine Aspiration of Gastric Contents | No Aspiration of Gastric Contents
Number analyzed (Participants) | 74 | 69
Hours | 402.6 [352.4 to 452.5] | 398.6 [350.3 to 447.0]
Statistical Analysis 1: Comparison: Routine Aspiration of Gastric Contents vs No Aspiration of Gastric Contents; Test type: Superiority; p = 0.95, Accelerated failure time regression mode

10. Secondary Outcome: Highest Alkaline Phosphatase Level
Description: Highest level during the first 42 days
Time Frame: baseline to 42 days
Measure: Median (Inter-Quartile Range); unit: Units/Liter
Arm/Group | Routine Aspiration of Gastric Contents | No Aspiration of Gastric Contents
Number analyzed (Participants) | 74 | 69
Units/Liter | 451 [371 to 664] | 495.5 [393 to 650.5]
Statistical Analysis 1: Comparison: Routine Aspiration of Gastric Contents vs No Aspiration of Gastric Contents; Test type: Superiority; p = 0.95, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: Occurrence of Cholestasis
Description: Occurrence of cholestatsis defined as a direct bilirubin level > 2 mg/dL
Time Frame: Baseline to 42 days
Measure: Least Squares Mean (95% Confidence Interval); unit: Events
Arm/Group | Routine Aspiration of Gastric Contents | No Aspiration of Gastric Contents
Number analyzed (Participants) | 74 | 69
Events | 0.040 [0.017 to 0.092] | 0.057 [0.025 to 0.131]
Statistical Analysis 1: Comparison: Routine Aspiration of Gastric Contents vs No Aspiration of Gastric Contents; Test type: Superiority; p = 0.23, Accelerated failure time regression mode

12. Secondary Outcome: Level of Direct Bilirubin
Description: Level of direct bilirubin on routine weekly or biweekly laboratory testing
Time Frame: Baseline to 42 days. highest value reported
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dl
Arm/Group | Routine Aspiration of Gastric Contents | No Aspiration of Gastric Contents
Number analyzed (Participants) | 74 | 69
mg/dl | 0.690 [0.568 to 0.819] | 0.671 [0.542 to 0.799]
Statistical Analysis 1: Comparison: Routine Aspiration of Gastric Contents vs No Aspiration of Gastric Contents; Test type: Superiority; p = 0.98, Mixed Models Analysis

13. Secondary Outcome: Length of Hospital Stay
Description: Days infant remains in hospital
Time Frame: baseline to approximately 3 months
Measure: Least Squares Mean (95% Confidence Interval); unit: days
Arm/Group | Routine Aspiration of Gastric Contents | No Aspiration of Gastric Contents
Number analyzed (Participants) | 74 | 69
days | 86.4 [80.7 to 92.1] | 79.1 [73.17 to 84.5]
Statistical Analysis 1: Comparison: Routine Aspiration of Gastric Contents vs No Aspiration of Gastric Contents; Test type: Superiority; p = 0.01, Accelerated failure time regression mode

14. Secondary Outcome: Episodes of Late Onset Sepsis
Description: Episodes of presumed or culture positive sepsis at > 3 days of life
Time Frame: 4 to 42 days
Measure: Least Squares Mean (95% Confidence Interval); unit: number of episodes
Arm/Group | Routine Aspiration of Gastric Contents | No Aspiration of Gastric Contents
Number analyzed (Participants) | 74 | 69
number of episodes | 1.38 [0.97 to 1.94] | 0.97 [0.67 to 1.40]
Statistical Analysis 1: Comparison: Routine Aspiration of Gastric Contents vs No Aspiration of Gastric Contents; Test type: Superiority; p = 0.08, Mixed Models Analysis

15. Secondary Outcome: Episodes of Necrotizing Enterocolitis
Description: Episodes of radiologic evidence of necrotizing enterocolitis (Stage 2 or greater)
Time Frame: Baseline to 42 days
Measure: Least Squares Mean (95% Confidence Interval); unit: number of episodes
Arm/Group | Routine Aspiration of Gastric Contents | No Aspiration of Gastric Contents
Number analyzed (Participants) | 74 | 69
number of episodes | 0.026 [0.006 to 0.109] | 0.008 [0.003 to 0.046]
Statistical Analysis 1: Comparison: Routine Aspiration of Gastric Contents vs No Aspiration of Gastric Contents; Test type: Superiority; p = 0.25, Mixed Models Analysis

16. Secondary Outcome: Episodes of Ventilator Associated Pneumonia
Description: Episodes of ventilator associated pneumonia
Time Frame: baseline to 42 days
Measure: Number; unit: episodes
Arm/Group | Routine Aspiration of Gastric Contents | No Aspiration of Gastric Contents
Number analyzed (Participants) | 74 | 69
episodes | 0 | 0

17. Secondary Outcome: Episodes of Aspiration Pneumonia
Description: Episodes of aspiration pneumonia on radiograph
Time Frame: baseline to 42 days
Measure: Median (Inter-Quartile Range); unit: episodes
Arm/Group | Routine Aspiration of Gastric Contents | No Aspiration of Gastric Contents
Number analyzed (Participants) | 74 | 69
episodes | 0 [0 to 0] | 0 [0 to 0]
Statistical Analysis 1: Comparison: Routine Aspiration of Gastric Contents vs No Aspiration of Gastric Contents; Test type: Superiority; p = 0.27, Wilcoxon (Mann-Whitney)

18. Secondary Outcome: Episodes of a Positive Tracheal Culture
Description: Episodes of a tracheal culture positive for bacteria
Time Frame: Baseline to 42 days
Measure: Least Squares Mean (95% Confidence Interval); unit: Episodes
Arm/Group | Routine Aspiration of Gastric Contents | No Aspiration of Gastric Contents
Number analyzed (Participants) | 74 | 69
Episodes | 0.055 [0.029 to 0.107] | 0.088 [0.058 to 0.152]
Statistical Analysis 1: Comparison: Routine Aspiration of Gastric Contents vs No Aspiration of Gastric Contents; Test type: Superiority; p = 0.17, Mixed Models Analysis

19. Secondary Outcome: Episodes of 2 or More Positive Tracheal Aspirate Cultures
Description: Episodes of 2 or more tracheal cultures positive for bacteria
Time Frame: Baseline to 42 days
Measure: Least Squares Mean (95% Confidence Interval); unit: episodes
Arm/Group | Routine Aspiration of Gastric Contents | No Aspiration of Gastric Contents
Number analyzed (Participants) | 74 | 69
episodes | 0.015 [0.007 to 0.033] | 0.024 [0.012 to 0.047]
Statistical Analysis 1: Comparison: Routine Aspiration of Gastric Contents vs No Aspiration of Gastric Contents; Test type: Superiority; p = 0.17, Mixed Models Analysis

20. Secondary Outcome: Episodes of Bronchopulmonary Dysplasia
Description: Episodes of bronchopulmonary dysplasia
Time Frame: Baseline to approximately 3 months
Measure: Least Squares Mean (95% Confidence Interval); unit: Episodes
Arm/Group | Routine Aspiration of Gastric Contents | No Aspiration of Gastric Contents
Number analyzed (Participants) | 74 | 69
Episodes | 0.512 [0.305 to 0.850] | 0.680 [0.414 to 1.12]
Statistical Analysis 1: Comparison: Routine Aspiration of Gastric Contents vs No Aspiration of Gastric Contents; Test type: Superiority; p = 0.43, Mixed Models Analysis

21. Secondary Outcome: Highest Tracheal Pepsin Level
Description: The highest level of pepsin obtained from endotracheal tube secretions
Time Frame: Baseline to 42 days
Measure: Median (Inter-Quartile Range); unit: ng/ml
Arm/Group | Routine Aspiration of Gastric Contents | No Aspiration of Gastric Contents
Number analyzed (Participants) | 74 | 69
ng/ml | 1 [0.2 to 5.71] | 0.9 [0 to 2]
Statistical Analysis 1: Comparison: Routine Aspiration of Gastric Contents vs No Aspiration of Gastric Contents; Test type: Superiority; p = 0.694, Wilcoxon (Mann-Whitney)

22. Secondary Outcome: Days of Invasive Ventilation
Description: Number of days infants required invasive ventilation
Time Frame: Baseline to approximately 3 months
Measure: Least Squares Mean (95% Confidence Interval); unit: days
Arm/Group | Routine Aspiration of Gastric Contents | No Aspiration of Gastric Contents
Number analyzed (Participants) | 74 | 69
days | 14.3 [11.2 to 17.4] | 13.3 [10.3 to 16.5]
Statistical Analysis 1: Comparison: Routine Aspiration of Gastric Contents vs No Aspiration of Gastric Contents; Test type: Superiority; p = 0.97, Accelerated failure time regression mode

23. Secondary Outcome: Number of Infants Who Died
Description: Number of infants who died during the 6 weeks study.
Time Frame: Baseline to 42 days
Measure: Number; unit: participants
Arm/Group | Routine Aspiration of Gastric Contents | No Aspiration of Gastric Contents
Number analyzed (Participants) | 74 | 69
participants | 6 | 1
Statistical Analysis 1: Comparison: Routine Aspiration of Gastric Contents vs No Aspiration of Gastric Contents; Test type: Superiority; p = 0.60, Mixed Models Analysis

24. Secondary Outcome: Number of Abdominal Radiographs
Description: number of abdominal radiographs performed
Time Frame: baseline to 42 days
Measure: Least Squares Mean (95% Confidence Interval); unit: number of episodes
Arm/Group | Routine Aspiration of Gastric Contents | No Aspiration of Gastric Contents
Number analyzed (Participants) | 74 | 69
number of episodes | 4.34 [3.66 to 5.34] | 3.81 [3.24 to 4.64]
Statistical Analysis 1: Comparison: Routine Aspiration of Gastric Contents vs No Aspiration of Gastric Contents; Test type: Superiority; p = 0.25, Mixed Models Analysis

25. Secondary Outcome: Episodes of Abdominal Distension
Description: Episodes of increased abdominal girth by 2cm or greater
Time Frame: Baseline to 42 days
Measure: Least Squares Mean (95% Confidence Interval); unit: episodes
Arm/Group | Routine Aspiration of Gastric Contents | No Aspiration of Gastric Contents
Number analyzed (Participants) | 74 | 69
episodes | 1.79 [1.27 to 2.53] | 0.590 [0.344 to 1.012]
Statistical Analysis 1: Comparison: Routine Aspiration of Gastric Contents vs No Aspiration of Gastric Contents; Test type: Superiority; p = 0.001, Mixed Models Analysis

26. Secondary Outcome: Emesis
Description: Number of emesis episodes
Time Frame: baseline to 42 days
Measure: Least Squares Mean (95% Confidence Interval); unit: episodes
Arm/Group | Routine Aspiration of Gastric Contents | No Aspiration of Gastric Contents
Number analyzed (Participants) | 74 | 69
episodes | 2.46 [1.70 to 3.56] | 5.01 [3.87 to 6.50]
Statistical Analysis 1: Comparison: Routine Aspiration of Gastric Contents vs No Aspiration of Gastric Contents; Test type: Superiority; p = 0.002, Mixed Models Analysis

27. Secondary Outcome: Weight
Description: Weight at 6 weeks of age. Note infants were born weighing < 1500 grams
Time Frame: 42 days
Measure: Least Squares Mean (95% Confidence Interval); unit: grams
Arm/Group | Routine Aspiration of Gastric Contents | No Aspiration of Gastric Contents
Number analyzed (Participants) | 74 | 69
grams | 1129.7 [1111 to 1148] | 1145 [1126 to 1164]
Statistical Analysis 1: Comparison: Routine Aspiration of Gastric Contents vs No Aspiration of Gastric Contents; Test type: Superiority; p = 0.03, Mixed Models Analysis

28. Secondary Outcome: Head Circumference
Description: Head circumference at 42 days
Time Frame: 42 days
Measure: Least Squares Mean (95% Confidence Interval); unit: centimeters
Arm/Group | Routine Aspiration of Gastric Contents | No Aspiration of Gastric Contents
Number analyzed (Participants) | 74 | 69
centimeters | 25.94 [25.71 to 26.17] | 25.85 [25.62 to 26.08]
Statistical Analysis 1: Comparison: Routine Aspiration of Gastric Contents vs No Aspiration of Gastric Contents; Test type: Superiority; p = 0.56, Mixed Models Analysis

29. Secondary Outcome: Length
Description: Length at 42 days
Time Frame: 42 days
Measure: Least Squares Mean (95% Confidence Interval); unit: centimeters
Arm/Group | Routine Aspiration of Gastric Contents | No Aspiration of Gastric Contents
Number analyzed (Participants) | 74 | 69
centimeters | 36.41 [36.08 to 36.74] | 36.78 [36.44 to 37.11]
Statistical Analysis 1: Comparison: Routine Aspiration of Gastric Contents vs No Aspiration of Gastric Contents; Test type: Superiority; p = 0.59, Mixed Models Analysis

30. Secondary Outcome: Presence of Blood in Stools
Description: Proportion of guaiac positive stools.
Time Frame: baseline to 42 days
Measure: Least Squares Mean (95% Confidence Interval); unit: proportion
Arm/Group | Routine Aspiration of Gastric Contents | No Aspiration of Gastric Contents
Number analyzed (Participants) | 74 | 69
proportion | 0.247 [0.203 to 0.290] | 0.254 [0.210 to 0.298]
Statistical Analysis 1: Comparison: Routine Aspiration of Gastric Contents vs No Aspiration of Gastric Contents; Test type: Superiority; p = 0.888, Mixed Models Analysis

31. Secondary Outcome: Level of Fecal Calprotectin
Description: Level of calprotectin in stools
Time Frame: 42 days
Measure: Least Squares Mean (95% Confidence Interval); unit: μg/g
Arm/Group | Routine Aspiration of Gastric Contents | No Aspiration of Gastric Contents
Number analyzed (Participants) | 61 | 63
μg/g | 557.8 [454.4 to 661.1] | 456.1 [353.7 to 558.5]
Statistical Analysis 1: Comparison: Routine Aspiration of Gastric Contents vs No Aspiration of Gastric Contents; Test type: Superiority; p = 0.694, Regression, Linear

32. Secondary Outcome: Serum Gastrin Level
Description: level of gastrin at 3 weeks
Time Frame: baseline to 21 days
Measure: Least Squares Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Routine Aspiration of Gastric Contents | No Aspiration of Gastric Contents
Number analyzed (Participants) | 54 | 53
pg/mL | 80.50 [62.59 to 98.41] | 92.29 [74.21 to 110.37]
Statistical Analysis 1: Comparison: Routine Aspiration of Gastric Contents vs No Aspiration of Gastric Contents; Test type: Superiority; p = 0.248, general linear mixed model

33. Secondary Outcome: Serum Motilin Level
Description: Serum motilin level at 21 days
Time Frame: baseline to 21 days
Measure: Least Squares Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Routine Aspiration of Gastric Contents | No Aspiration of Gastric Contents
Number analyzed (Participants) | 50 | 55
pg/mL | 228.5 [191.8 to 265.1] | 225.8 [180.6 to 262.1]
Statistical Analysis 1: Comparison: Routine Aspiration of Gastric Contents vs No Aspiration of Gastric Contents; Test type: Superiority; p = 0.694, general linear mixed model

34. Secondary Outcome: Fecal S100A12
Description: Level of fecal S100A12
Time Frame: 42 days
Measure: Least Squares Mean (95% Confidence Interval); unit: ng/g
Arm/Group | Routine Aspiration of Gastric Contents | No Aspiration of Gastric Contents
Number analyzed (Participants) | 61 | 63
ng/g | 195.2 [119.2 to 271] | 144.4 [68.9 to 220]
Statistical Analysis 1: Comparison: Routine Aspiration of Gastric Contents vs No Aspiration of Gastric Contents; Test type: Superiority; p = 0.195, Regression, Linear

ADVERSE EVENTS:
Time Frame: 42 days
Arm/Group | Routine Aspiration of Gastric Contents | No Aspiration of Gastric Contents
All-Cause Mortality (participants affected / at risk) | 6/74 | 1/69
Serious Adverse Events (participants affected / at risk) | 7/74 | 8/69
Other Adverse Events (participants affected / at risk) | 0/74 | 0/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Routine Aspiration of Gastric Contents (N=74) | No Aspiration of Gastric Contents (N=69)
necrotizing enterocolits or spontaneous intestinal perforation (Gastrointestinal disorders) | 7 (7) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form: Protocol, statistical analysis and ICF (2016-03-04): https://cdn.clinicaltrials.gov/large-docs/43/NCT01863043/Prot_SAP_ICF_000.pdf